CLINICAL TRIAL: NCT03870529
Title: A Pilot Study of Neoadjuvant High Dose Vitamin A for Resectable Non-Small Cell Lung Cancer
Brief Title: High Dose Vitamin A Compound in Treating Participants With Resectable Non-Small Cell Lung Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00050640; NCI-2018-00888 (Other: Clinical Trial Reporting Program); WFBCCC 62218 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer; Stage I Lung Cancer; Stage Ib Lung Carcinoma; Stage IA Lung Carcinoma AJCC V7; Stage IIA Lung Carcinoma; Stage IIIA Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Vitamin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin A compound (Experimental): Participants receive vitamin A compound PO for 7 consecutive days in the absence of disease progression or unacceptable toxicity. Within 21 days of completing treatment, participants then undergo surgical resection.
  Interventions: Drug: Vitamin A Compound
- Therapeutic Conventional Surgery (Active Comparator): Description Participants undergo surgical resection.
  Interventions: Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Vitamin A Compound — Participants randomized to this arm will receive 7 consecutive days of of Vitamin A compound without disease progression or unacceptable toxicities. Within 21 days of completion of treatment participants will undergo surgical resection
  Other Names: Dimethyl-9-(2,6,6-trimethyl-1-cyclohexen-1-yl)-2,4,6,8-nonatetraen-1-ol, 68-26-8, A 313, Anti-Infective Vitamin, Anti-Infective vitamin, Antixerophthalmic Vitamin, Antixerophthalmic vitamin
  Arms: Vitamin A compound
Procedure: Therapeutic Conventional Surgery — Participants randomized to this arm will receive surgical resection
  Arms: Therapeutic Conventional Surgery

SUMMARY:
This trial studies how well high dose vitamin A compound works in treating participants with non-small cell lung cancer that can be removed by surgery. Vitamin A compound may increase the number of germinal centers (immune centers that make antibodies mature) in tumor and lymph tissues which may be beneficial to patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the percentage of resected cancers containing germinal centers (GCs) in patients who receive neoadjuvant vitamin A compound (vitamin A) to controls.

SECONDARY OBJECTIVES:

I. To compare the abundance of GCs in adjacent lymph nodes in patients who receive neoadjuvant vitamin A to controls.

II. To compare histopathologic responses based on tumor necrosis in lung cancer patients who receive neoadjuvant vitamin A to controls.

III. To compare overall survival of patients who receive neoadjuvant vitamin A to controls.

EXPLORATORY OBJECTIVES:

I. To describe immunophenotypic changes of monocytes including myeloid derived suppressor cells (MDSCs) in pre- and post-treatment blood samples.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive vitamin A compound orally (PO) for 7 consecutive days in the absence of disease progression or unacceptable toxicity. Within 21 days of completing treatment, participants then undergo surgical resection.

GROUP II: Participants undergo surgical resection.

After completion of study treatment, participants are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patients must have either biopsy proven or radiographically suspected non-small cell lung cancer.
* Patients must have disease in the chest that is felt to be surgically resectable.
* ECOG performance status of 0-2.
* Ability to understand and the willingness to sign an IRB-approved informed consent document

Exclusion Criteria:

* Patients younger than 18 years of age
* Women who are pregnant or breast feeding.
* Patients may not be receiving any other investigational agents for the treatment of nonsmall cell lung cancer.
* Patients may not be taking the following medications: high dose vitamin A supplement (multivitamin supplements prohibited only if vitamin A content is greater than 3,500 international units), bexarotene, alitretinoin, tretinoin, adapalene, isotretinoin, acitretin, doxycycline, minocycline, or demeclocycline,
* Uncontrolled intercurrent illness including, but not limited to, pancreatitis, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Hypervitaminosis A - toxic effects of ingesting too much vitamin A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Petty, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (9.0) | 69.1 (10.8) | 67.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Presence or Absence of Germinal Centers in Resected Tissue
Description: Presence/absence of germinal centers (GCs) in resected cancer tissues from patients who receive neoadjuvant vitamin A and controls.
Time Frame: Up to 2 years
Population: No samples were analyzed for outcomes and the study was stopped therefore data was not collected for outcome measures
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Germinal Centers in Lymph Nodes
Description: Measurement of GCs per unit area in adjacent lymph nodes will be assessed using semi-quantitative designation (Score of high, moderate, low, or absent) in patients who receive neoadjuvant vitamin A and controls.
Time Frame: Up to 2 years
Population: No samples were analyzed for outcomes and the study was stopped therefore data was not collected for outcome measures
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Presence or Absence of Tumor Necrosis
Description: Pathologic response will be defined by tumor necrosis which will be dichotomized as present or absent in patients who receive neoadjuvant vitamin A and controls
Time Frame: Up to 2 years
Population: No samples were analyzed for outcomes and the study was stopped therefore data was not collected for outcome measures
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival of patients receiving neoadjuvant Vitamin A and in controls.
Time Frame: Up to 2 years
Population: No samples were analyzed for outcomes and the study was stopped therefore data was not collected for outcome measures
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after last dose of study drug is administered
Arm/Group | Vitamin A Compound | Therapeutic Conventional Surgery
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03870529/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03870529/ICF_002.pdf